CLINICAL TRIAL: NCT01532037
Title: A Randomised Controlled Trial of Cognitive Behavioural Therapy Based Self Help for Fatigue in Multiple Sclerosis
Brief Title: Self Help for Fatigue in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RCT-MS-NHS-1
Record Dates: First submitted 2012-01-17; First posted 2012-02-13 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: Randomised controlled trial; Multiple Sclerosis; Fatigue; Cognitive Behavioural Therapy; Self Help
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Guided Self Help (Experimental): Participant receives usual care and 4, 45 minute sessions with a therapist to support them to complete the cognitive behavioural therapy based workbook for fatigue in Multiple Sclerosis.
  Interventions: Other: Cognitive behavioural therapy based self help
- Pure Self Help (Experimental): Participant receives usual care and cognitive behavioural therapy based self help work book for fatigue in multiple sclerosis to complete alone
  Interventions: Other: Cognitive behavioural therapy based self help
- Treatment as Usual (Placebo Comparator): Participants receive usual care from healthcare professionals
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Cognitive behavioural therapy based self help — Comparison of cognitive behavioural therapy based pure self help and guided self help (support of a therapist) compared to treatment as usual
  Arms: Guided Self Help; Pure Self Help
Other: Treatment as usual — Usual care from healthcare professionals with regard to patients symptoms of fatigue
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to determine if cognitive behavioural therapy (CBT) based self help is effective for the management of symptoms of fatigue in Multiple Sclerosis (MS).

DETAILED DESCRIPTION:
Background: Fatigue is a common disabling symptom in patients with Multiple Sclerosis (MS). Cognitive behavioural therapy (CBT) has been shown to be effective in the reduction of fatigue in MS and CBT-based self-help has been shown to be effective as a low intensity intervention for anxiety and depression.

Objectives: To evaluate the effectiveness of a CBT based self-help workbook at reducing perceived impact of fatigue in a clinical sample of MS patients.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be aged 18 or over
* Will have a recognised diagnosis of relapsing remitting or primary progressive relapsing remitting Multiple Sclerosis from a neurologist
* Cognitively able to give informed consent as deemed by referring clinician in the Fife Rehabilitation Service
* Willing to consent to randomised control trial
* Fatigue as a primary symptom

Exclusion Criteria:

* Patients with severe anxiety or depression (assessed by cut off on HADS)
* Patients with psychosis or personality disorders (assessed by referring clinician)
* Patients currently receiving input from psychological services for fatigue management
* Patients with suicidal ideation or plans (assessed by referring clinician)
* Patients who are unable to read the workbook or standardised questionnaires due to literacy levels or cognitive abilities will be excluded from the analysis, although if patients have literacy or cognitive problems, referral to a more suitable 1-to-1 type of therapy will be made.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline on ratings of the Modified Fatigue Impact Scale at post measure, 3, 6 & 12 months follow up. | 5 time points at 0, 8, 20, 32 & 60 weeks.
  The Modified Fatigue Impact Scale (MFIS) consists of 21 items selected from the Fatigue Impact Scale (FIS; Fisk, Ritvo, Ross, Haase, Murray, & Schlech, 1994), a multidimensional scale developed to assess the perceived impact of fatigue on a variety of daily activities. The items of the MFIS can be combined into three subscales (Physical, Cognitive, and Psychosocial), as well as into a total MFIS score. All items are scaled so that higher scores indicate a greater impact of fatigue on a patient's activities. Measures will be taken at 5 time points to assess change over time.

SECONDARY OUTCOMES:
Change from baseline on the 36-Item Short Form Survey Instrument at post measure, 3, 6 and 12 months follow up. | 5 time points at 0, 8, 20, 32 & 60 weeks
  36-Item Short Form Survey Instrument (SF 36, Ware et al.1993) consists of 36 questions measuring functional health and well-being from the patient's point of view. Scores are split into two summary measures (physical health and mental health) and within the two summary measures there are eight scales which include. The eight scales are made up of; physical functioning, role limitations due to physical functioning, bodily pain, general health, vitality, social functioning, role limitations due to emotional functioning and mental health.
Change from baseline on the Hospital Anxiety and Depression Scale at post measure, 3, 6 and 12 months follow up. | 5 time points at 0, 8, 20, 32 & 60 weeks
Change from baseline on the Self-Efficacy for managing chronic Disease 6 Item Scale at post measure, 3, 6 and 12 months follow up. | 5 time points at 0, 8, 20, 32 & 60 weeks
  Is a 6-item scale which is adapted from the original 33 item scale (Lorig et al. 1996). The 6-item scale was developed so it would be less burdensome for patients. The 6- item scale covers areas of symptom control, role function, emotional functioning and communicating with physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Nesbitt, Principal Investigator — National Health Service, University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Fife Rehabilitation Service, Leven, Scotland
  - NHS Fife, Leven, Scotland

REFERENCES:
- [Result] Chapter 4 in https://era.ed.ac.uk/bitstream/handle/1842/21011/Gallen2015.pdf